CLINICAL TRIAL: NCT04758117
Title: Real-World Effectiveness of Upadacitinib in Patients Joining Subgroups Either With Oligo- or Poly-ArtIcular Psoriatic Arthritis on Minimal Disease Activity
Brief Title: A Study to Assess the Change in Disease State in Adult Participants Being Treated With Oral Upadacitinib Tablets in Participants With Oligo- or Poly-artIcular Psoriatic Arthritis
Acronym: UPJOINT
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-483
Record Dates: First submitted 2021-02-16; First posted 2021-02-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; Oligoarticular Psoriatic Arthritis; Polyarticular Psoriatic Arthritis; Upadacitinib; Rinvoq
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants Receiving Upadacitinib: Participants receiving Upadacitinib for psoriatic arthritis (PsA).

SUMMARY:
Psoriatic arthritis (PsA) is a type of arthritis (swelling and stiffness in the joints) that is frequently seen in trial participants who also have the skin condition psoriasis. It is caused by the body's immune system mistakenly attacking healthy joint tissue causing inflammation, joint damage, disability, and a reduced life expectancy. The main objective of this study is to characterize attainment of minimal disease activity (MDA) at week 24 under continuous treatment with upadacitinib in participants with oligo- or polyarticular PsA as part of real-world practice.

Upadacitinib is a drug approved for the treatment of Psoriatic arthritis (PsA) in Germany and Canada. Approximately 380 adult participants with PsA at multiple sites in Germany and Canada.

Participants will receive oral Upadacitinib tablets per current local label, according to local standard of care and international guidelines.

There may be a higher burden for participants in this study compared to standard of care. Participants will attend regular visits per routine clinical practice. The effect of the treatment will be checked by medical assessments, checking for side effects, and by questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of active Psoriatic Arthritis (PsA) upon judgment of the treating physician.
* Swollen joint count (SJC) >= 1 out of 66 joints.
* Decision on the treatment with Upadacitinib was made prior to any decision to approach the participant to participate in this study.

Exclusion Criteria:

* Cannot be treated with Upadacitinib according to the local Upadacitinib Summary of Product Characteristics (SmPC).
* Prior treatment with Upadacitinib.
* Currently participating in interventional research or within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with psoriatic arthritis (PsA).
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Receiving Upadacitinib who Attain Minimal Disease Activity (MDA) | At Week 24
  MDA will be determined based on participants fulfilling 5 of 7 outcome measures: tender joint count 68 (TJC68) <= 1, swollen joint count (SJC66) ≤ 1, body surface area (BSA) <= 3%; Patient's Assessment of Pain numeric rating scale (NRS) <= 1.5, Patient's Global Assessment of Disease Activity (PtGA) NRS <= 2.0, Health Assessment Questionnaire Disability Index (HAQ-DI) <= 0.5, tender entheseal points <= 1.

SECONDARY OUTCOMES:
Percentage of Participants Maintaining MDA Under Upadacitinib Treatment, in Participants who had Achieved MDA at Week 24 | At Week 48
  MDA will be determined based on participants fulfilling 5 of 7 outcome measures: TJC68 <= 1, SJC66 ≤ 1, BSA <= 3%; Patient's Assessment of Pain NRS <= 1.5, PtGA NRS <= 2.0, HAQ-DI <= 0.5, tender entheseal points <= 1.
Mean change in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Question 2 (Pain in Neck, Back or Hip) | Baseline to Week 48
  The BASDAI consists of a 0 - 10 scale measuring discomfort, pain, and fatigue (0 being no problem and 10 being the worst problem).
Mean Change in Disease Activity in PSoriatic Arthritis score (DAPSA) | Baseline to Week 48
  The DAPSA is a numerical sum of the 66 swollen and 68 tender joint counts, the participant pain and global assessments (each on a 0-10 scale) and C-reactive protein (CRP) (in mg/dL), thus ranging from 0 to about 160.
Mean Change in Percentage of Participants with Dactylitis | Baseline to Week 48
  Mean change in percentage of participants with dactylitis.
Mean Change in Number of Fingernails Affected with Psoriasis | Baseline to Week 48
  Mean change in number of fingernails affected with psoriasis.
Mean Change in 12-Item Short Form Health Survey (SF-12) | Baseline to Week 48
  The SF-12 is a 12-item, patient-reported, generic, non-disease specific, overall HRQoL instrument with extensive use in multiple disease states.
Mean Change in Dermatology Life Quality Index (DLQI) [in Participants with Skin Involvement] | Baseline to Week 48
  The DLQI consists of 10 questions concerning participants' perception of the impact of the skin disease on different aspects of their HRQoL over the previous week.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (93):
- Canada (18):
  - Dr. Jonathan D. Chan Inc. /ID# 241611, Vancouver, British Columbia
  - Manitoba Clinic /ID# 234148, Winnipeg, Manitoba
  - The Waterside Clinic /ID# 234146, Barrie, Ontario
  - Dr. Chrisostomos Kouroukis & Dr. Pauline Boulos MPC /ID# 233565, Dundas, Ontario
  - Arthur Karasik Medicine Professional Corporation /ID# 234147, Etobicoke, Ontario
  - Lau Bacchus Professional Medicine Corp /ID# 245283, Hamilton, Ontario
  - Credit Valley Rheumatology /ID# 234144, Mississauga, Ontario
  - Dr. L. Lisnevskaia Medicine Professional Corporation /ID# 239611, Oshawa, Ontario
  - Angela Montgomery Medicine Professional Corporation /ID# 239608, Ottawa, Ontario
  - Niagara Peninsula Arthritis Ct /ID# 245521, St. Catharines, Ontario
  - Dr. Sabeen Anwar Medicine Professional Corporation /ID# 242696, Windsor, Ontario
  - Applied Medical Informatics Research Inc. (AMIR) /ID# 239614, Montreal, Quebec
  - Clinique de Rhumatologie de Montreal /ID# 239613, Montreal, Quebec
  - CISSSBSL -Hopital regional de Rimouski /ID# 234150, Rimouski, Quebec
  - Groupe de Recherche en Maladies Osseuses Inc /ID# 234145, Sainte-Foy, Quebec
  - CIUSSS de l'Estrie - CHUS /ID# 241054, Sherbrooke, Quebec
  - Centre de Recherche Musculo-Squelettique /ID# 234151, Trois-Rivières, Quebec
  - Dr Naik-Medical Professional Corporation-Alliance Health /ID# 234149, Saskatoon, Saskatchewan
- Germany (75):
  - Praxis Dr. Rinaldi /ID# 228639, Ulm, Baden-Wurttemberg
  - Praxis Dres. Kellerer/Kellerer/Krüger /ID# 227414, Munich, Bavaria
  - Rheumahaus Studien GbR, Potsdam, DE /ID# 230771, Potsdam, Brandenburg
  - Internistisches Praxiszentrum /ID# 228262, Giessen, Hesse
  - Fachpraxis fuer Rheumatologie und Osteologie /ID# 227391, Bruchhausen-Vilsen, Lower Saxony
  - Kupka & Kupka, Altenburg, DE /ID# 228243, Altenburg
  - Marycz, Amberg, DE /ID# 227413, Amberg
  - Rheumapraxis am Webereck /ID# 229274, Augsburg
  - MVZ Weserbergland /ID# 228806, Bad Pyrmont
  - ACURA Rheumazentrum Baden-Bade /ID# 239202, Baden-Baden
  - Rheumapraxis Prof Dr Karin Manger /ID# 229120, Bamberg
  - Sozialstiftung Bamberg /ID# 228549, Bamberg
  - Internistische-rheumatologische Praxisgemeinschaft /ID# 228240, Bayreuth
  - MVZ Rheumatologie /ID# 240868, Berlin
  - Praxis Dr. med. Angela Seifert /ID# 233772, Berlin
  - Praxis Dr. Silke Zinke /ID# 229127, Berlin
  - Rheumapraxis am Schlachtensee /ID# 228800, Berlin
  - Eisterhues, Braunschweig, DE /ID# 227390, Braunschweig
  - Dres. Schuh /ID# 227411, Coburg
  - Rheumatologie in Veedel /ID# 228469, Cologne
  - Krankenhaus Porz am Rhein /ID# 228358, Cologne
  - Praxis Dr. Kirrstetter /ID# 229609, Deggendorf
  - Kreiskrankenhaus Demmin /ID# 228253, Demmin
  - Rheumatologisches MVZ Dresden /ID# 230787, Dresden
  - Praxis Dilltal /ID# 228640, Ehringshausen
  - MVZ Ambulantes Rheumazentrum Erfurt /ID# 248933, Erfurt
  - Dres. Waehrisch/Flaxenberg /ID# 228263, Essen
  - Michael Mueller, Freiberg, DE /ID# 228468, Freiberg
  - Praxis Dr. Behringer /ID# 229275, Fulda
  - Rockwitz, Goslar, DE /ID# 227856, Goslar
  - Praxis Fiene /ID# 244732, Greifswald
  - Praxis Dr. Kuehne /ID# 229119, Haldensleben I
  - Praxis Dr. Liebhaber /ID# 228636, Halle
  - Stille, Hanover, DE /ID# 229604, Hanover
  - Heilig, Heidelberg, DE /ID# 228356, Heidelberg
  - St. Elisabeth Gruppe GmbH -Katholische Kliniken /ID# 228797, Herne
  - Praxis Bernd Mueller /ID# 230776, Homburg
  - Praxis K. Pagel /ID# 228247, Hoppegarten
  - Kremers, Juelich, DE /ID# 240383, Jülich
  - Rheumapraxis Kaufering /ID# 231391, Kaufering
  - Alb-Donau Klinikum, Langenau /ID# 233770, Langenau
  - Hamann & Teich & Boche,Leipzig /ID# 228355, Leipzig
  - Praxis internistische Rheumatologie /ID# 227857, Leipzig
  - Dres. Teipel/Toussaint/Saech /ID# 228465, Leverkusen
  - Dr. Bolze, Ludwigshafen, DE /ID# 230773, Ludwigshafen
  - Aurich & Sieburg, Magdeburg /ID# 229605, Magdeburg
  - Praxis Dr. Annekatrin Rossbach /ID# 230783, Mansfeld / Großörner
  - Harmuth, Marktredwitz, DE /ID# 227709, Marktredwitz
  - RHIO Forschungsinstitut /ID# 227736, Meerbusch
  - Vollmer & Partner, DE /ID# 240869, Mönchengladbach
  - Prof-med-stud.de /ID# 228637, Munich
  - Rheumatologische Facharztpraxis /ID# 228808, Naumburg
  - Berger, Naunhof, DE /ID# 229612, Naunhof
  - Praxis Dr. med Thilo Klopsch /ID# 229123, Neubrandenburg
  - Erbsloeh-Moeller, Neunkirchen /ID# 230778, Neunkirchen
  - MVZ Medic-Center Nürnberg GmbH /ID# 240982, Nuremberg
  - Die Fachaerzte im Rottal - Nephrologie, Rheumatologie /ID# 230774, Pfarrkirchen
  - MVZ für Rheumatologie Dr. M. Welcker /ID# 227858, Planegg
  - Baumann & Lang, Plauen, DE /ID# 229128, Plauen
  - Praxis Dr. Sabine Reckert /ID# 248986, Potsdam
  - Knappschaftsklinikum Saar /ID# 248882, Püttlingen
  - Rheumazentrum Ratingen /ID# 228261, Ratingen
  - Rheumatologische Praxis Dr. Jochen Walter /ID# 229607, Rendsburg
  - Rheumatologische Gemeinschaftspraxis Schwerin /ID# 228260, Schwerin
  - Melzer, Seesen, DE /ID# 227386, Seesen
  - Barmherzige Bruder MVZ Klinikum Straubing GmbH /ID# 228805, Straubing
  - Krankenhaus der Barmherzigen Brueder Trier /ID# 229603, Trier
  - Praxis Dr. Haas /ID# 228813, Tübingen
  - Rheumathologie Ulm /ID# 238801, Ulm
  - MVZ Lahn-Dill-Kliniken GmbH /ID# 231390, Wetzlar
  - MVZ Lahn-Dill-Kliniken GmbH /ID# 262011, Wetzlar
  - Krankenhaus St. Josef /ID# 229611, Wuppertal
  - Praxis Barmen /ID# 227392, Wuppertal
  - Sprekeler, Zeven, DE /ID# 233773, Zeven
  - Fricke-Wagner, Zwickau, DE /ID# 230775, Zwickau

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Werner SG, Schwarze I, Baraliakos X, Fiene M, Walter J, Girard T, Laliberte MC, Jeromin K, Baschuk N, Allard-Charmard H, Bessette L, Hueber AJ. Effectiveness and Safety of Upadacitinib in Treating Oligoarticular and Polyarticular Psoriatic Arthritis: Primary Analysis from the UPJOINT-Study. Rheumatol Ther. 2026 Feb;13(1):45-64. doi: 10.1007/s40744-025-00802-5. Epub 2025 Nov 5. PMID 41191276
- [Derived] Werner SG, Baraliakos X, Reckert S, Bohl-Buhler M, Laliberte MC, Girard T, Jeromin K, Baschuk N, Fritz B, Bessette L, Hueber AJ. Treatment with Upadacitinib in Active Psoriatic Arthritis: Efficacy and Safety Data of the First 192 Patients from the UPJOINT Study, a Multicentre, Observational Study in Clinical Practice. Rheumatol Ther. 2023 Dec;10(6):1503-1518. doi: 10.1007/s40744-023-00589-3. Epub 2023 Sep 11. PMID 37695506
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P20-483#additional-resources-section